CLINICAL TRIAL: NCT04115501
Title: Intraoperative Fraction of Inspired Oxygen and Lung Injury in Coronary Artery Bypass Grafting Surgery
Brief Title: Intra-operative Fraction of Inspired Oxygen and Lung Injury in Coronary Artery Bypass Grafting Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to enroll
Sponsor: University of Louisville (Other)
Collaborators: Peking Union Medical College Hospital (Other); Tianjin Chest Hospital (Other); Xiangya Hospital of Central South University (Other); Guangdong Provincial People's Hospital (Other); Second Xiangya Hospital of Central South University (Other); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jiapeng Huang, Principal Investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19.0988
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Lung Injury; Pulmonary Complication
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research fellows and ICU physicians who record and assess the primary and secondary outcomes will be blinded to the group assignment. The principal investigator (PI) of every center and the physicians who conduct the anesthesia and monitoring intraoperatively in operating room are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive Oxygen (Experimental): The restrictive oxygen patients' Fraction of Inspired Oxygen (FiO2) will be set at a minimum of 0.3 to maintain their oxygen saturations (SpO2) greater than or equal to 95% intraoperatively. During CPB a blended air/oxygen mixture will be titrated to arterial blood gas analysis with aim of maintenance of PaO2 between 100 and 150 mmHg. After transfer to ICU, all patients' FiO2 will be set to 50% initially, and titrate to minimal FiO2 (not less than 21%) for maintain SPO2≥95% until extubation.
  Interventions: Other: Fraction of Inspired Oxygen
- Liberal Oxygen (No Intervention): The liberal oxygen group will consist of subjects exposed to a Fraction of Inspired Oxygen (FiO2) set at 1.0 throughout the intraoperative period, including during cardiopulmonary bypass. After transfer to ICU, all patients' FiO2 will be set to 50% initially, and titrate to minimal FiO2 (not less than 21%) for maintain SPO2≥95% until extubation.

INTERVENTIONS:
Other: Fraction of Inspired Oxygen — Fraction of Inspired Oxygen during cardiac surgery, including cardiopulmonary bypass
  Arms: Restrictive Oxygen

SUMMARY:
This study is a prospective observer blinded, central randomization controlled, multi-center clinical trial to assess the relationship between intraoperative FiO2 and postoperative pulmonary complications with lung injury.

DETAILED DESCRIPTION:
Hyperoxia is common in cardiac surgery and is easy to prevent by adjusting FiO2. Since there is no prospective study on different FiO2 and postoperative pulmonary complications (PPCs) during cardiac surgery. We hypothesized that hyperoxia during cardiac surgery could lead to higher incidence of lung injury and PPCs than normoxia. The objective of this trial is to compare postoperative PPCs and other outcomes between hyperoxia and normoxia strategy by PaO2/FiO2 in CABG patients.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75
* BMI from 20 to 39.9
* ASA II/III
* Undergoing isolated selective on-pump CABG through median sternotomy
* Subsequent admission to an intensive care unit (ICU).

Exclusion Criteria:

* with severe chronic obstructive pulmonary disease (COPD)
* Pregnant woman.
* With current acute coronary syndrome (<1 week)
* Severe anemia (hemoglobin <10g/L)
* Preoperative supplemental oxygen requirement to maintain arterial O2 of 92%,
* Right to left shunt in heart
* Carotid stenosis defined as >50% stenosis of either carotid artery,
* Cardiac surgery that requires intraoperative circulatory arrest,
* Current use of dialysis,
* One-lung ventilation during surgery,
* Recent smoking (within 1 month),
* Non-respiratory reason to reintubate or delayed extubation such as bleeding or heart failure,
* Perioperative allogenic transfusion with red blood cell, plasma or platelet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-27 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
arterial PO2/FiO2 Ratio | 48hr post operation
  minimal postoperative arterial PO2/FiO2 Ratio

SECONDARY OUTCOMES:
Pulmonary complications | up to one week while in the hospital
  ARDS, noncardiogenic pulmonary edema, pulmonary infection, pneumonia, pleural effusion, atelectasis, and respiratory failure are secondary endpoints
length of mechanical ventilation | up to one week while in the hospital
  time from skin closure to extubation
length of postoperative ICU stay | up to one week while in the hospital
  time from ICU entry to discharge from ICU
length of hospital stay | up to one week while in the hospital
  time from surgery day to discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Jiapeng Huang, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No